CLINICAL TRIAL: NCT05382065
Title: The Correlation Between Period of Anemia and Duration of Mechanical Ventilation in Patients Admitted to the Surgical Intensive Care Unit
Brief Title: Anemia and Duration of Mechanical Ventilation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Annop Piriyapatsom, MD, Associate Professor, Mahidol University
Other Study IDs: 255/2565(IRB3)
Record Dates: First submitted 2022-05-16; First posted 2022-05-19 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Anemia; Mechanical Ventilation; Critically Ill; Intensive Care Unit; Morality; Organ Dysfunction Syndrome
Keywords: Duration of mechanical ventilation; Duration of anemia; Intensive care unit; Mortality; Organ dysfunction
MeSH Terms: conditions — Anemia; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In mechanically ventilated patients in intensive care unit, anemia is commonly seen and it is probably associated with adverse outcomes including mortality. We aim to investigate the impact of duration of anemia and the duration of mechanical ventilation as well as clinical outcomes in critically ill patients in intensive care unit who required ventilatory support >96 hr.

DETAILED DESCRIPTION:
Anemia is one of the most common conditions encountered critically ill patients. Various mechanisms can put these patients at risk of anemia including gastrointestinal hemorrhage, iron deficiency, inflammation and infection, stress, and multiple blood testing. Anemia can affect cardiopulmonary function as depletion in oxygen content in body. In mechanically ventilated patients, anemia is associated with increased duration of mechanical ventilation, increased length of stay, and possibly increased mortality. Some research suggested that hemoglobin level <8.5 g/dl was a potential risk factor for adverse outcome in critically ill patients required mechanical ventilation >96 hr. However, most researches focused on hemoglobin levels and the associated adverse events in mechanically ventilated patients. To the best of our knowledge, there are few studies reported the impact of the duration of anemia and the clinical outcomes in these patients. We hypothesize that the short duration of anemia developed in mechanically ventilated patients has no effect on duration of mechanical ventilation. We, therefore, aim to investigate the impact of the duration of anemia on duration of mechanical ventilation in critically ill patients required ventilatory support >96 hours.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose age of equal or more than 18 years old
* Patients admitted to the surgical intensive care unit during the study period
* Patients required ventilatory support with invasive mechanical ventilation for more than 96 hours

Exclusion Criteria:

* Patients whose data regarding time of beginning or ending of ventilatory support missed
* Patients who are previously included in this study and are re-admitted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to the surgical intensive care unit and required ventilatory support with invasive mechanical ventilation for more than 96 hours
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-07-08 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Duration of mechanical ventilation | 28 days after initiation of ventilatory support
  Days patients received mechanical ventilation

SECONDARY OUTCOMES:
Duration of anemia | 28 days after initiation of ventilatory support
  Days patients had hemoglobin level <8 g/dl while they were on ventilatory support
Cardiovascular dysfunction | 28 days after initiation of ventilatory support
  SOFA cardiovascular component equal to 1, 3, or 4
Respiratory dysfunction | 28 days after initiation of ventilatory support
  SOFA respiratory component >1
Renal dysfunction | 28 days after initiation of ventilatory support
  SOFA respiratory component >1
Gastrointestinal dysfunction | 28 days after initiation of ventilatory support
  SOFA gastrointestinal component >1
Hematologic dysfunction | 28 days after initiation of ventilatory support
  SOFA hematologic component >1
ICU length of stay | Up to 90 days following inclusion
  Duration from ICU admission to ICU discharge
Hospital length of stay | Up to 90 days following inclusion
  Duration from hospital admission to hospital discharge
ICU mortality | Up to 90 days following inclusion
  Status at ICU discharge either alive or deceased
Hospital mortality | Up to 90 days following inclusion
  Status at hospital discharge either alive or deceased

CONTACTS AND LOCATIONS:
Overall Officials: Annop Piriyapatsom, MD, Principal Investigator — Department of Anesthesiology, Faculty of Medicine Siriraj Hospital, Mahidol University
Locations (1):
- Department of Anesthesiology, Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok Noi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hebert PC, Blajchman MA, Cook DJ, Yetisir E, Wells G, Marshall J, Schweitzer I; Transfusion Requirements in Critical Care Investigators for the Canadian Critical Care Trials Group. Do blood transfusions improve outcomes related to mechanical ventilation? Chest. 2001 Jun;119(6):1850-7. doi: 10.1378/chest.119.6.1850. PMID 11399714
- [Background] Hayden SJ, Albert TJ, Watkins TR, Swenson ER. Anemia in critical illness: insights into etiology, consequences, and management. Am J Respir Crit Care Med. 2012 May 15;185(10):1049-57. doi: 10.1164/rccm.201110-1915CI. Epub 2012 Jan 26. PMID 22281832
- [Background] Zilberberg MD, Stern LS, Wiederkehr DP, Doyle JJ, Shorr AF. Anemia, transfusions and hospital outcomes among critically ill patients on prolonged acute mechanical ventilation: a retrospective cohort study. Crit Care. 2008;12(2):R60. doi: 10.1186/cc6885. Epub 2008 Apr 28. PMID 18442375
- [Background] Penuelas O, Frutos-Vivar F, Fernandez C, Anzueto A, Epstein SK, Apezteguia C, Gonzalez M, Nin N, Raymondos K, Tomicic V, Desmery P, Arabi Y, Pelosi P, Kuiper M, Jibaja M, Matamis D, Ferguson ND, Esteban A; Ventila Group. Characteristics and outcomes of ventilated patients according to time to liberation from mechanical ventilation. Am J Respir Crit Care Med. 2011 Aug 15;184(4):430-7. doi: 10.1164/rccm.201011-1887OC. PMID 21616997
- [Background] Zilberberg MD, Luippold RS, Sulsky S, Shorr AF. Prolonged acute mechanical ventilation, hospital resource utilization, and mortality in the United States. Crit Care Med. 2008 Mar;36(3):724-30. doi: 10.1097/CCM.0B013E31816536F7. PMID 18209667
- [Background] Ghiani A, Sainis A, Sainis G, Neurohr C. Anemia and red blood cell transfusion practice in prolonged mechanically ventilated patients admitted to a specialized weaning center: an observational study. BMC Pulm Med. 2019 Dec 18;19(1):250. doi: 10.1186/s12890-019-1009-1. PMID 31852456
- [Background] Mueller MM, Van Remoortel H, Meybohm P, Aranko K, Aubron C, Burger R, Carson JL, Cichutek K, De Buck E, Devine D, Fergusson D, Follea G, French C, Frey KP, Gammon R, Levy JH, Murphy MF, Ozier Y, Pavenski K, So-Osman C, Tiberghien P, Volmink J, Waters JH, Wood EM, Seifried E; ICC PBM Frankfurt 2018 Group. Patient Blood Management: Recommendations From the 2018 Frankfurt Consensus Conference. JAMA. 2019 Mar 12;321(10):983-997. doi: 10.1001/jama.2019.0554. PMID 30860564
- [Background] Hebert PC, Wells G, Blajchman MA, Marshall J, Martin C, Pagliarello G, Tweeddale M, Schweitzer I, Yetisir E. A multicenter, randomized, controlled clinical trial of transfusion requirements in critical care. Transfusion Requirements in Critical Care Investigators, Canadian Critical Care Trials Group. N Engl J Med. 1999 Feb 11;340(6):409-17. doi: 10.1056/NEJM199902113400601. PMID 9971864
- [Background] Vlaar AP, Oczkowski S, de Bruin S, Wijnberge M, Antonelli M, Aubron C, Aries P, Duranteau J, Juffermans NP, Meier J, Murphy GJ, Abbasciano R, Muller M, Shah A, Perner A, Rygaard S, Walsh TS, Guyatt G, Dionne JC, Cecconi M. Transfusion strategies in non-bleeding critically ill adults: a clinical practice guideline from the European Society of Intensive Care Medicine. Intensive Care Med. 2020 Apr;46(4):673-696. doi: 10.1007/s00134-019-05884-8. Epub 2020 Jan 7. PMID 31912207
- [Background] Lai YC, Ruan SY, Huang CT, Kuo PH, Yu CJ. Hemoglobin levels and weaning outcome of mechanical ventilation in difficult-to-wean patients: a retrospective cohort study. PLoS One. 2013 Aug 28;8(8):e73743. doi: 10.1371/journal.pone.0073743. eCollection 2013. PMID 24015310